CLINICAL TRIAL: NCT01731002
Title: A Phase 2, Double-masked, Randomized, Multi-center, Active-controlled, Dose-response Parallel-group Study Comparing the Safety and Ocular Hypotensive Efficacy of AR-13324 to Latanoprost in Patients With Elevated Intraocular Pressure
Brief Title: Study Comparing the Safety and Efficacy of AR-13324 to Latanoprost in Patients With Elevated Intraocular Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AR-13324-CS202
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2016-06

CONDITIONS: Ocular Hypertension; Open Angle Glaucoma
Keywords: Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle; Glaucoma | interventions — netarsudil; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AR-13324 Ophthalmic Solution 0.01% (Experimental): 1 drop to study eye once daily
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.01%
- AR-13324 Ophthalmic Solution 0.02% (Experimental): 1 drop to study eye once daily
  Interventions: Drug: AR-13324 Ophthalmic Solution 0.02%
- Latanoprost Ophthalmic Solution 0.005% (Active Comparator): 1 drop to study eye once daily
  Interventions: Drug: Latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: AR-13324 Ophthalmic Solution 0.01% — Administered to study eye, once daily (QD) in the evening (PM) for 28 days
  Arms: AR-13324 Ophthalmic Solution 0.01%
Drug: AR-13324 Ophthalmic Solution 0.02% — Administered to study eye, QD in the PM for 28 days
  Other Names: Netarsudil
  Arms: AR-13324 Ophthalmic Solution 0.02%
Drug: Latanoprost ophthalmic solution 0.005% — Administered to study eye, QD in the PM for 28 days
  Other Names: Latanoprost
  Arms: Latanoprost Ophthalmic Solution 0.005%

SUMMARY:
Double-masked, randomized, multi-center, dose-response, active-controlled parallel-comparison of AR-13324 to latanoprost

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or greater.
2. Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT).
3. Unmedicated (post-washout) Intraocular Pressure (IOP) ≥ 24 mm Hg at 2 eligibility visits (08:00 hr), 2-7 days a part, and ≥ 22 mm Hg at 10:00 and 16:00 hrs at the second qualification visit. If only one eye meets the IOP criteria it must be the same eye that met the criteria at all the qualification timepoints.
4. Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200).
5. Able and willing to give signed informed consent and follow study instructions.

Exclusion Criteria:

Ophthalmic

1. Glaucoma: pseudoexfoliation or pigment dispersion component, history of angle closure or narrow angles. Note: Previous laser peripheral iridotomy is NOT acceptable.
2. IOP > 36 mm Hg.
3. Known hypersensitivity to any component of the formulation (benzalkonium chloride, etc.), or to topical anesthetics.
4. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s, e.g., laser trabeculoplasty).
5. Refractive surgery in study eye(s) (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser eye surgery (LASIK), etc.).
6. Ocular trauma within the past six months, or ocular surgery or laser treatment within the past three months prior to screening.
7. Evidence of ocular infection, inflammation, clinically significant blepharitis or conjunctivitis at screening (Visit 0), or a history of herpes simplex keratitis
8. Ocular medication of any kind within 30 days of Visit 0, with the exception of a) ocular hypotensive medications (which must be washed out according to the provided schedule), b) lid scrubs (which may be used prior to, but not after Visit 0) or c) lubricating drops for dry eye (which may be used throughout the study).
9. Clinically significant ocular disease (e.g. uveitis, severe keratoconjunctivitis sicca) which might interfere with the study, including glaucomatous damage so severe that washout of ocular hypotensive medications for one month is not judged safe (i.e., cup-disc ratio > 0.8).
10. Central corneal thickness greater than 600 µm.
11. Any abnormality preventing reliable applanation tonometry of either eye.

    Systemic:
12. Clinically significant abnormalities (as determined by the treating physician) in laboratory tests at screening.
13. Known hypersensitivity or contraindication to latanoprost.
14. Clinically significant systemic disease (e.g., myasthenia gravis, hepatic, renal, endocrine or cardiovascular disorders) which might interfere with the study.
15. Participation in any investigational study within 30 days prior to screening.
16. Changes of systemic medication that could have a substantial effect on IOP within 30 days prior to screening, or anticipated during the study.
17. Due to the current status of the preclinical safety program, women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the screening examination and must not intend to become pregnant during the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Heah, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (22):
- United States (22):
  - Kenneth Sall, M.D., Artesia, California
  - United Medical Research Institute, Inglewood, California
  - Aesthetic Eye Care Institute, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Centre For Health Care, Poway, California
  - Clayton Eye Center, Morrow, Georgia
  - Coastal Research Associates, LLC, Roswell, Georgia
  - Bradley Kwapiszeski, MD, Shawnee Mission, Kansas
  - Taustine Eye Center, Louisville, Kentucky
  - Alan L Robin, M.D., Baltimore, Maryland
  - Seidenberg Protzko Eye Associates, Havre de Grace, Maryland
  - Great Lakes Eye Care, Saint Joseph, Michigan
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Rochester Ophthalmological Group, Rochester, New York
  - Charlotte Eye Ear Nose and Throat, Charlotte, North Carolina
  - Michael E. Tepedino, M.D., High Point, North Carolina
  - The Eye Institute, Tulsa, Oklahoma
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Texan Eye, Austin, Texas
  - Cataract & Glaucoma Center, El Paso, Texas
  - Medical Center Ophth. Associates, San Antonio, Texas
  - Virginia Eye Consultants, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- AR-13324 Ophthalmic Solution 0.01%; AR-13324 Ophthalmic Solution 0.02%; Latanoprost Ophthalmic Solution 0.005%: 1 drop to study eye once daily (QD) in the evening (PM)
Period: Overall Study
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Started | 75 | 72 | 77
Completed | 71 | 68 | 74
Not Completed | 4 | 4 | 3
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Non-Compliant | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Test Agent Discontinuation | 0 | 1 | 0
Not completed — Uncontrolled Intraocular Pressure (IOP) | 2 | 0 | 0
Not completed — Elevated IOP | 1 | 0 | 0
Not completed — Inappropriate use of study medications | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005% | Total
Number analyzed (Participants) | 75 | 72 | 77 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.54) | 66.3 (10.25) | 65.7 (11.82) | 65.1 (11.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 45 | 132
  Male | 33 | 27 | 32 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 15 | 46
  Not Hispanic or Latino | 59 | 57 | 62 | 178
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 16 | 19 | 52
  White | 56 | 53 | 58 | 167
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: The primary efficacy endpoint was the mean IOP across subjects within treatment group on each day at each post-treatment timepoint. IOP was measured at 0800, 1000, and 1600 hours on days 0, 14, and 28. IOP was also measured at 0800 hours on Day 7 and follow-up days 29 and 30.
Time Frame: Study treatment was administered for 28 days
Population: Modified intent to treat (mITT) population (3 subjects were excluded, leaving 221)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 74 | 71 | 76
mmHg
  Day 0, 0800 hours | 27.34 (3.529) | 27.11 (3.031) | 26.78 (2.749)
  Day 0, 1000 hours | 25.55 (3.411) | 25.41 (3.024) | 25.18 (2.719)
  Day 0, 1600 hours | 24.49 (3.128) | 24.29 (2.602) | 24.58 (2.515)
  Day 7, 0800 hours | 21.89 (4.672) | 21.15 (4.047) | 20.03 (3.173)
  Day 14, 0800 hours | 21.24 (4.295) | 20.80 (3.679) | 19.30 (3.033)
  Day 14, 1000 hours | 19.28 (3.581) | 18.88 (3.461) | 18.09 (2.884)
  Day 14, 1600 hours | 18.90 (3.578) | 18.72 (3.585) | 17.86 (2.977)
  Day 28, 0800 hours | 21.95 (4.717) | 21.24 (4.034) | 19.24 (2.899)
  Day 28, 1000 hours | 19.69 (4.358) | 19.53 (3.726) | 18.40 (2.994)
  Day 28, 1600 hours | 18.82 (3.281) | 19.13 (3.656) | 18.34 (3.052)

2. Secondary Outcome: Extent of Exposure
Description: Exposure to study medication in days for all treatment groups.
Time Frame: 28 Days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
Number analyzed (Participants) | 75 | 72 | 77
days | 27.6 (4.07) | 26.8 (4.6) | 27.8 (1.35)

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | AR-13324 Ophthalmic Solution 0.01% | AR-13324 Ophthalmic Solution 0.02% | Latanoprost Ophthalmic Solution 0.005%
All-Cause Mortality (participants affected / at risk) | 1/75 | 0/72 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/75 | 0/72 | 2/77
Other Adverse Events (participants affected / at risk) | 43/75 | 45/72 | 18/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.01% (N=75) | AR-13324 Ophthalmic Solution 0.02% (N=72) | Latanoprost Ophthalmic Solution 0.005% (N=77)
Pneumonia Streptococcal (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR-13324 Ophthalmic Solution 0.01% (N=75) | AR-13324 Ophthalmic Solution 0.02% (N=72) | Latanoprost Ophthalmic Solution 0.005% (N=77)
Conjunctival Hyperaemia (Eye disorders) | 29 | 34 | 12
Ocular Hyperaemia (Eye disorders) | 10 | 7 | 0
Lacrimation Increased (Eye disorders) | 4 | 5 | 0
Conjunctival Haemorrhage (Eye disorders) | 4 | 4 | 0
Foreign Body Sensation in Eyes (Eye disorders) | 0 | 5 | 3
Instillation Site Pain (General disorders) | 5 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No